CLINICAL TRIAL: NCT02008201
Title: Vitamin D Status and Supplementation in Elite Athletes
Brief Title: Vitamin D Status and Supplementation in Athletes
Acronym: D-status
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Wageningen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D-status
Record Dates: First submitted 2013-09-10; First posted 2013-12-11 (Estimated); Last update posted 2014-12-15 (Estimated); Status verified 2013-12

CONDITIONS: Vitamin D Deficiency
Keywords: dose-response study
MeSH Terms: conditions — Vitamin D Deficiency | interventions — Vitamin D

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Vitamin D dose 1 (Experimental): Vitamin D dose 1
  Interventions: Dietary Supplement: vitamin D
- Vitamin D dose 2 (Experimental): Vitamin D dose 2
  Interventions: Dietary Supplement: vitamin D
- Vitamin D dose 3 (Experimental): Vitamin D dose 3
  Interventions: Dietary Supplement: vitamin D
- observational (No Intervention): No dose

INTERVENTIONS:
Dietary Supplement: vitamin D
  Arms: Vitamin D dose 1; Vitamin D dose 2; Vitamin D dose 3

SUMMARY:
The objectives of this study are 1) to assess the prevalence of vitamin D deficiency in a group of sub elite athletes and 2) to identify seasonal changes in vitamin D status and the effect that supplementation may have during the course of a year.

The study is a double blinded parallel study design.

DETAILED DESCRIPTION:
Study population: 175 elite/ sub elite athletes, male and female, aged 18-60y, from a variety of sport disciplines

ELIGIBILITY:
Inclusion Criteria:

* athletes
* 19-60y

Exclusion Criteria:

* subjects who take vitamin D supplements

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 153 (Actual)
Dates: Start 2012-05; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Change in serum 25(OH)D | Every 3 months during one year

CONTACTS AND LOCATIONS:
Overall Officials: Lisette de Groot, Prof. Dr., Principal Investigator — Wageningen University
Locations (1):
- Wageningen University, Wageningen, Netherlands